CLINICAL TRIAL: NCT00162305
Title: A Double-blind, Placebo-controlled, Randomized, Multiple-dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Bms-512148 in Diabetic Subjects
Brief Title: A Phase IIA Study of BMS-512148 to Assess Safety, Exposure, and Biological Effects in Stable Type 2 Diabetic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-003
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: BMS-512148
- 2 (Active Comparator)
  Interventions: Drug: BMS-512148
- 3 (Active Comparator)
  Interventions: Drug: BMS-512148
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-512148 — Capsules, Oral, 100 mg, Once daily, 14 days.
  Other Names: Dapagliflozin
  Arms: 1
Drug: BMS-512148 — Capsules, Oral, 25 mg, Once daily, 14 days.
  Other Names: Dapagliflozin
  Arms: 2
Drug: BMS-512148 — Capsules, Oral, 5 mg, Once daily, 14 days.
  Other Names: Dapagliflozin
  Arms: 3
Drug: Placebo — Capsules, Oral, 0 mg, Once daily, 14 days.
  Other Names: Dapagliflozin
  Arms: 4

SUMMARY:
The purpose of this clinical research study is to assess the safety of, exposure to, and biological effects of BMS-512148 in stable Type 2 diabetic subjects

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Type 2 diabetes mellitus, who are treated with metformin or diet alone (drug naive).
* Fasting glucose (FG) < - 240 mg/dL, while on metformin or antidiabetic diet alone.
* HbA1c (Hemoglobin A1c) in the range of 6.0-10.0%

Exclusion Criteria:

* Women of childbearing potential

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple oral doses of BMS-512148 administered alone or concomitantly with metformin in diabetic subjects | 14 days
  Adverse event monitoring, physical examinations, clinical laboratory determinations, electrocardiograms (ECG), and vital sign assessments

SECONDARY OUTCOMES:
To assess the PK of BMS-512148 and its pharmacologically active metabolite, BMS-511926, when BMS-512148 is administered alone or concomitantly with metformin | 14 days
  Exposure to BMS-512148 and BMS-511926
To assess the pharmacodynamic effect of BMS-512148, administered alone or concomitantly with metformin, on serum and urine markers of glucose homeostasis | 14 days
  Fasting and post-prandial serum glucose, serum fructosamine, serum insulin, and serum C-peptide and urinary glucose and urinary calcium
To assess the effect of BMS-512148, administered alone or concomitantly with metformin, on safety markers in urine | 14 days
  calcium, magnesium, sodium, potassium, phosphate, chloride, uric acid, oxalate, citrate, total protein, albumin, osmolality, deoxypyridinoline (D-pyr) cross-links, C-telopetide (CTX), N-acetyl-β- D-glucoasaminidase (NAG), and β2-microglubulin (β2-MG)
To assess the effect of BMS-512148, administered alone or concomitantly with metformin, on the following safety markers in serum | 14 days
  Serum osteocalcin, parathyroid hormone (PTH), 25-Vitamin D, and 1,25-Vitamin D
To assess the effect of BMS-512148 administered alone or concomitantly with metformin on the percent inhibition of renal glucose reabsorption | 14 days
  Percent inhibition of renal glucose resorption over each 0-4 h, 4-8 h, and 8-12 h post-dose interval calculated from the amount of renally filtered glucose and the amount of glucose excreted in the urine for each collection interval.
To assess the effects of BMS-512148 on the PK of metformin in diabetic subjects. | 14 days
  Exposure to metformin
To identify potential biomarkers in both urine and blood | 14 days
  Serum and urine for metabonomic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, New Orleans, Louisiana
  - Local Institution, San Antonio, Texas

REFERENCES:
- [Result] Komoroski B, Vachharajani N, Feng Y, Li L, Kornhauser D, Pfister M. Dapagliflozin, a novel, selective SGLT2 inhibitor, improved glycemic control over 2 weeks in patients with type 2 diabetes mellitus. Clin Pharmacol Ther. 2009 May;85(5):513-9. doi: 10.1038/clpt.2008.250. Epub 2009 Jan 7. PMID 19129749
- See also: MB102-003 _CSR_synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3630&filename=MB102-003%20_CSR_synopsis.pdf